CLINICAL TRIAL: NCT03145636
Title: The ReNEW Study: Maestro® New Enrollment Post-Approval Study Protocol
Acronym: ReNEW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D01569-000
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Obesity, Morbid
Keywords: Obesity; Bariatric surgery; Vagal blocking; vBloc therapy; Vagus Nerve; Percent excess weight loss; Percent total body weight loss
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Observational arm (Other): Subjects will receive the device implant and use the vBloc Achieve Weight Management Program.
  Interventions: Device: vBloc Maestro Rechargeable System; Other: vBloc Achieve Weight Management Program
- Randomized sub-study -Treatment (Other): Subjects will be randomly assigned (1:1) either to treatment or control. Treatment arm will receive the device and use of vBloc Achieve Weight Management Program.
  Interventions: Device: vBloc Maestro Rechargeable System; Other: vBloc Achieve Weight Management Program
- Randomized sub-study - Control (Other): Subjects will be randomly assigned (1:1) either to treatment or control. Control will participate in a Control Weight Management (CWM) program for 6 months prior to receiving the device implant and using the vBloc Achieve program.
  Interventions: Device: vBloc Maestro Rechargeable System; Other: vBloc Achieve Weight Management Program; Other: Control Weight Management (CWM) program

INTERVENTIONS:
Device: vBloc Maestro Rechargeable System — Intra-abdominal vagal blocking neuromodulation device for the treatment of obesity
Other: vBloc Achieve Weight Management Program — Remotely accessible web-based program to add additional support to subjects with vBloc therapy
Other: Control Weight Management (CWM) program — In person visits with Registered Dietician, or trained staff who will counsel subjects on energy balance, dietary intake, physical activity and eating behavior modification.
  Arms: Randomized sub-study - Control

SUMMARY:
This is a five-year, single arm, multi-center trial to evaluate the long-term safety and efficacy of the Maestro Rechargeable System in treating obesity. The study will include an observational arm and a randomized sub-study.

DETAILED DESCRIPTION:
The study evaluates the safety and efficacy of the vBloc Therapy delivered by the Maestro Rechargeable System for the treatment obesity. The Maestro Rechargeable System delivers intermittent, electrical blocking signals to the anterior and posterior trunks of the intra-abdominal vagus nerve (termed vBloc Therapy) and is designed to reduce sensations of hunger and produce satiety leading to weight loss.

Subjects in the observational arm (100 subjects total) will receive the device implant and use the vBloc Achieve Weight Management Program.

The randomized sub-study (100 subjects) will randomly assign subjects (1:1) to either treatment (50 subjects) or control (50 subjects). The treatment arm will receive the device implant and use of the vBloc Achieve Weight Management Program. The control arm will participate in the Control Weight Management (CWM) during a 6 month period prior to receiving the device implant and using the vBloc Achieve program.

The vBloc Achieve Weight Management Program consists of recommendations regarding diet, exercise and behavior modification, and will be utilized by all subjects following their device implant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Body mass index (BMI) ≥ 40 kg/m2 to 45 kg/m2 or BMI ≥ 35 kg/m2 to 39.9 kg/m2 with one or more obesity related co-morbid conditions
3. Females or males. Note: females of child-bearing potential must have a negative urine pregnancy test at Screen and also within 14 days of implant procedure followed by physician-approved contraceptive regimen for the duration of the study period.
4. At least 18 years of age
5. Failure to respond to supervised diet/exercise program(s) in which the subject was engaged within the last five years
6. Ability to complete all study visits and procedures

Exclusion Criteria:

1. Patients with cirrhosis of the liver, portal hypertension, or esophageal varices.
2. Patients with a large (>5cm) symptomatic hiatal hernia
3. Patients for whom magnetic resonance imaging (MRI) is planned
4. Patients at high risk for surgical complications
5. Patients who have a permanently implanted, electrical-powered medical device or gastrointestinal device or prosthesis (e.g. pacemakers, implanted defibrillators, neurostimulators)
6. Patients for whom shortwave, microwave, or therapeutic ultrasound diathermy is planned Note: Diathermy is any treatment that uses high-frequency electromagnetic radiation, electric currents, or ultrasonic waves to produce heat in body tissues. Patients absolutely CANNOT be treated with any type of shortwave, microwave, or therapeutic ultrasound diathermy device whether or not it is used to produce heat. These treatments should not be applied anywhere on the body.
7. Current medical condition that, in the opinion of the investigator, would make the subject unfit for surgery or that would be exacerbated by intentional weight loss. Some examples include diagnosis of cancer, recent heart attack, recent stroke or serious trauma.
8. Recent cessation of cigarette smoking (prior 2 months)
9. History of bariatric surgery, Nissen fundoplication, gastric resection, major upper-abdominal surgery, or other abdominal procedures at the discretion of the investigator (acceptable surgeries include cholecystectomy or hysterectomy)
10. Patients with recent (<2 years) or current history of illicit drug abuse
11. Patients with significant psychiatric disease including borderline personality disorder, psychosis, schizophrenia, unstable depression, suicidal ideation, or mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of device, therapy and procedure-related serious adverse events (SAEs) | 5 years
  The primary safety objective is to show that the rate of serious adverse events (SAEs) related to the device, implant/revision procedure (including explant procedure), general surgical procedure, or therapy algorithm is statistically lower than 25% at 5 years.

OTHER OUTCOMES:
Rate of therapy-related adverse events at 5 years | 5 years
  To evaluate the long-term (5-year) rate of therapy-related adverse events
Rate of device-related malfunction at 5 years | 5 years
  To evaluate the long-term (5-year) rate of device (neuroregulator or lead) malfunction requiring a revision procedure
Mean percentage excess weight loss (%EWL) through 5 years | 5 years
  To evaluate the mean percentage excess weight loss (%EWL) through 5 years
Percentage of subjects achieving at least 20 and 25%EWL thresholds through 5 years | 5 years
  To evaluate the percentage of subjects achieving at least 20% EWL and 25% EWL through 5 years
Mean percentage total body weight loss (%TBL) through 5 years | 5 years
  To evaluate the mean percentage total body weight loss (%TBL) through 5 years
Mean percentage of subjects achieving at least 5 and 10% TBL through 5 years | 5 years
  To evaluate the percentage of subjects achieving at least 5% TBL and 10% TBL through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Billington, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - HonorHealth, Scottsdale, Arizona
  - Winthrop University Hospital, Mineola, New York

IPD SHARING:
Plan to Share IPD: No